CLINICAL TRIAL: NCT06704581
Title: A Multicenter, Randomized, Double-blind, Placebo-parallel Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of BGM0504 Injection in Chinese Non-diabetes Participants with Overweight or Obese
Brief Title: A Study of BGM0504 Injection in Participants with Obesity or Overweight
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BrightGene New Bio-Medical Technology(Wuxi) Co.Ltd. (Industry)
Responsible Party: Sponsor
Organization: BrightGene Bio-Medical Technology Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGM0504-Ⅲ-WL
Record Dates: First submitted 2024-11-07; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 5 mg BGM0504 injection (Experimental)
  Interventions: Drug: 5 mg BGM0504 injection
- 10 mg BGM0504 injection (Experimental)
  Interventions: Drug: 10 mg BGM0504 injection administered subcutaneously (SC) once a week
- 15 mg BGM0504 injection (Experimental)
  Interventions: Drug: 15 mg BGM0504 injection
- BGM0504 placebo (Placebo Comparator)
  Interventions: Drug: BGM0504 placebo

INTERVENTIONS:
Drug: 5 mg BGM0504 injection — 5mg BGM0504 injection administered subcutaneously (SC) once a week.
  Arms: 5 mg BGM0504 injection
Drug: 10 mg BGM0504 injection administered subcutaneously (SC) once a week — 10mg BGM0504 injection administered subcutaneously (SC) once a week.
  Arms: 10 mg BGM0504 injection
Drug: 15 mg BGM0504 injection — 15mg BGM0504 injection administered subcutaneously (SC) once a week.
  Arms: 15 mg BGM0504 injection
Drug: BGM0504 placebo — BGM0504 placebo administered SC once a week.
  Arms: BGM0504 placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase III validation clinical study in Chinese adult non-diabetic overweight or obese Participants. The main purpose is to evaluate the clinical efficacy of BGM0504 injection for 36 weeks of administration as an adjunct to diet, exercise, and behavioral interventions in overweight or obese non-diabetic adults in China for weight management, and to evaluate the clinical efficacy and safety of BGM0504 injection for 52 weeks of administration.

ELIGIBILITY:
Inclusion Criteria:

* A male or female aged 18 to 65 years inclusive at screening
* BMI≥28 kg/m², or 24.0≤BMI<28.0 kg/m² and previous diagnosis with at least one of the following comorbidities: i. Prediabetes (impaired fasting blood glucose and/or impaired glucose tolerance), hypertension, nonalcoholic fatty liver disease, or one or more of these; ii. Joint pain with weight bearing; iii. Dyspnea caused by obesity or obstructive sleep apnea syndrome
* Weight change < 5.0% (chief complaint) after diet and exercise control for at least 12 weeks before screening
* Female participants who are not pregnant or lactating. Female participants with childbearing potential and their partners should use highly effective, medically accepted contraception, will not have pregnancy and fertility plan, and refrain from donating ovum until one month after the end of the study

Exclusion Criteria:

* Diabetes mellitus
* Known to be allergic to 3 or more kinds of foods or medications, or allergic to GLP-1 agonist, or have a severe allergic disease (asthma, urticaria, eczematous dermatitis, etc.) at screening
* Has been treated with GLP-1 receptor agonists or similar drugs containing the same target, or drugs used for weight control in the three months prior to screening
* Secondary disease or drug-induced obesity, including : elevated cortisol (e.g. Cushing's syndrome), obesity due to pituitary and hypothalamic damage, obesity due to diet drug reduction/discontinuation, etc.;
* History of pancreatitis
* Have the currently uncontrolled thyroid diseases with stable treatment dose and clinically significant abnormal results of thyroid function test occurred at screening
* Previous history of moderate or severe depression, or PHQ-9 score ≥15, or history of other serious mental illness, or Any lifetime history of a suicide attempt

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-11-27 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline,Week 36
  Change from baseline in body weight after 36 weeks of treatment
Percentage of Participants Who Achieve≥5% Body Weight Reduction | Baseline,Week 36
  Percentage of Participants Who Achieve≥5% Body Weight Reduction

SECONDARY OUTCOMES:
Percent Change From Baseline in Body Weight | Baseline, Week 52
  Percent Change from Baseline in Body Weight after 52weeks of treatment
Change From Baseline in Body Weight | Baseline, Week36 and 52
  Change from baseline in body weight
Percentage of Participants Who Achieve≥5% Body Weight Reduction | Baseline, Week 36 and 52
  Percentage of Participants Who Achieve≥5% Body Weight Reduction
Percentage of Participants Who Achieve≥10% Body Weight Reduction | Baseline, Week 36 and 52
  Percentage of Participants Who Achieve≥10% Body Weight Reduction
Percentage of Participants Who Achieve≥15%Body Weight Reduction | Baseline, Week 36 and 52
  Percentage of Participants Who Achieve≥15%Body Weight Reduction
Percentage of Participants Who Achieve≥20% Body Weight Reduction | Baseline, Week 36 and 52
  Percentage of Participants Who Achieve≥20% Body Weight Reduction.
Change From Baseline in Waist Circumference | Baseline, Week 36 and 52
  Change From Baseline in Waist Circumference after 52weeks of treatment.
Change From Baseline in Body Mass Index (BMI) | Baseline, Week 36 and 52
  Change From Baseline in Body Mass Index (BMI) after 52weeks of treatment
Change From Baseline in Fasting Glucose | Baseline, Week 36 and 52
  Change From Baseline in Fasting Glucose after 52weeks of treatment
Change From Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 36 and 52
  Change From Baseline in Hemoglobin A1c (HbA1c) after 52weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China